CLINICAL TRIAL: NCT03850574
Title: A Phase 1/2 Open Label, Multicenter, Dose Escalation and Expansion Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HM43239 in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Tuspetinib (HM43239) in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Acronym: TUSCANY
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aptose Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HM-FLTI-101; 2023-503244-14-00 (EU CTIS Number); 2022-002826-29 (EudraCT Number)
Record Dates: First submitted 2019-01-28; First posted 2019-02-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Leukemia, Myeloid, Acute; Refractory AML; Relapsed Adult AML; Myelodysplastic Syndrome With Excess Blasts-2; Chronic Myelomonocytic Leukemia
Keywords: Tuspetinib; Acute Myeloid Leukemia; AML; Relapsed; Refractory; Myelodysplastic Syndromes with Increased Blasts Grade 2; MDS-IB2; Chronic Myelomonocytic Leukemia; CMML; Venetoclax; Azacitidine; Newly Diagnosed
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Recurrence | interventions — venetoclax; Azacitidine; Infusions, Intravenous

STUDY DESIGN:
Intervention Model Description: 1. Part A: Tuspetinib dose escalation
  2. Part B: Tuspetinib dose exploration
  3. Part C: Tuspetinib monotherapy dose expansion
  4. Part C: Tuspetinib in combination with venetoclax ("doublet" therapy) dose expansion
  5. Part D: Tuspetinib in combination with venetoclax and azacitidine ("triplet" therapy) dose exploration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part A Dose Escalation [COMPLETED] (Experimental): Part A dose escalation of tuspetinib as a single agent is planned for up to 6 dose levels. If a study participant in dose escalation at any dose level achieves clinical response, then the dose level will continue to enroll in Part B. If one DLT or less is observed in the 6 participants (<1/6 DLT observed) in Part A, up to 20 evaluable participants can be enrolled in Part B at that dose level.
  Interventions: Drug: Tuspetinib
- Part B Dose Exploration [ACTIVE, NOT RECRUITING] (Experimental): Part B dose exploration of tuspetinib as a single agent is planned for up to 4 dose levels.
  Interventions: Drug: Tuspetinib
- Part C Dose Expansion (tuspetinib as a single agent) [COMPLETE] (Experimental): Part C dose expansion of tuspetinib as a single agent is planned for 2 dose levels. Study participants will be randomly assigned to either arm based on the number of slots available. The initial tuspetinib dose will be 120 mg.
  Interventions: Drug: Tuspetinib
- Part C Dose Expansion (tuspetinib plus venetoclax) [COMPLETE] (Experimental): Part C dose expansion of tuspetinib in combination with venetoclax is planned for 2 dose levels. The initial tuspetinib dose will be 80 mg.
  Interventions: Drug: Tuspetinib; Drug: Venetoclax Oral Tablet
- Part D Dose Exploration (tuspetinib plus venetoclax and azacitidine) [ACTIVE, RECRUITING - US Sites] (Experimental): Part D dose exploration of tuspetinib in combination with venetoclax and azacitidine is planned for up to 6 dose levels. The initial tuspetinib dose will be 40 mg.
  Interventions: Drug: Tuspetinib; Drug: Venetoclax Oral Tablet; Drug: Azacitidine for Intravenous Infusion

INTERVENTIONS:
Drug: Tuspetinib — Daily (QD), continuous dosing
  Other Names: HM43239
Drug: Venetoclax Oral Tablet — Venetoclax will be given to study participants in the Part C tuspetinib plus venetoclax combination treatment group either in 50 mg or 100 mg tablets
  Other Names: Venetoclax
  Arms: Part C Dose Expansion (tuspetinib plus venetoclax) [COMPLETE]; Part D Dose Exploration (tuspetinib plus venetoclax and azacitidine) [ACTIVE, RECRUITING - US Sites]
Drug: Azacitidine for Intravenous Infusion — Azacitidine will be given to study participants in Part D as intravenous infusion at a dose of 75 mg/m^2
  Other Names: Azacitidine
  Arms: Part D Dose Exploration (tuspetinib plus venetoclax and azacitidine) [ACTIVE, RECRUITING - US Sites]

SUMMARY:
The main purpose of this study is to identify a safe and potentially effective dose of tuspetinib to be used in future studies in study participants diagnosed with acute myeloid leukemia (AML), myelodysplastic syndromes with increased blasts grade 2 (MDS-IB2), or chronic myelomonocytic leukemia (CMML) that is relapsed or refractory after at least one line of prior therapy, or in study participants with newly diagnosed AML. Tuspetinib will be administered as a single agent or in combination with other drugs (venetoclax or venetoclax plus azacitidine), as specified for each part of the study.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, multi-center study designed to assess the efficacy, safety, tolerability, and pharmacokinetics, including determining the recommended Phase 2 dose (RP2D) of tuspetinib (HM43239) in subjects with relapsed or treatment-refractory acute myeloid leukemia (AML).

Part C: This portion of the study will evaluate tuspetinib (HM43239) as monotherapy in patients with relapsed or refractory (R/R) AML, focusing on safety, tolerability, pharmacokinetics, and preliminary efficacy (Aptivate).

Part D: This portion of the study will evaluate the safety, tolerability, and PK parameters of tuspetinib (HM43239) in combination with venetoclax and azacitidine when administered to newly diagnosed AML patients who are ineligible for induction chemotherapy (Tuscany).

ELIGIBILITY:
Inclusion Criteria for Parts A/B/C:

* Study participant is defined as having morphologically documented primary or secondary AML, MDS-IB2 (≥ 10% bone marrow blasts), or CMML by the World Health Organization (WHO) criteria (2016), and fulfills one of the following:

  1. Refractory to at least 1 cycle of prior therapy
  2. Relapsed after achieving remission with a prior therapy
* Study participant has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Study participant's interval from prior treatment to time of study drug administration is at least 2 weeks for cytotoxic agents (except hydroxyurea given for controlling blast cells), at 4 weeks for biologic or cellular immunotherapies, or least 5 half-lives for prior experimental agents or noncytotoxic agents, including immunosuppressive therapy post hematopoietic stem cell transplantation (HSCT). Upon discussion with the Medical Monitor, a shorter than stated washout period may be considered provided that the study participant has recovered from any clinically relevant safety issue and recovered to Grade ≤ 1 toxicity from prior therapies.
* Study participant must meet the following criteria as indicated on the clinical laboratory tests.

  1. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3× institutional upper limit normal (ULN)
  2. Total serum bilirubin ≤ 1.5× institutional ULN
  3. Creatinine clearance as calculated by the Cockcroft-Gault formula or measured by 24-h urine collection of > 45 mL/min.
* Study participant is suitable for oral administration of study drug and has minimum life expectancy (≥ 3 months)
* Female study participants must be either:
* Of non-childbearing potential

  1. Post-menopausal (defined as at least 1 year without any menses) prior to screening, or
  2. Documented surgically sterile or status post hysterectomy (at least 1 month prior to screening)
* Or, if of childbearing potential,

  1. Must have a negative serum or urine pregnancy test at screening (within 72 hours prior to start of treatment), and
  2. Must use an acceptable highly effective method of birth control starting at screening and throughout the study period and for 90 days after the final study drug administration.
* Female study participants must not be breastfeeding at screening and during the study period, and for 90 days after the final study drug administration
* Female study participants must not donate ova starting at screening and throughout the study period, and for 90 days after the final study drug administration.
* Male study participants and their female spouse/partners who are of childbearing potential must be using highly effective contraception starting at screening and continue throughout the study period and for 90 days after the final study drug administration.
* Male study participants must not donate sperm starting at screening and throughout the study period and for 90 days after the final study drug administration.
* Study participant agrees not to participate in another interventional study while on treatment.

Exclusion Criteria for Parts A/B/C:

Study participants must not enter the study if any of the following exclusion criteria are met:

* Study participant was diagnosed with acute promyelocytic leukemia (APL).
* Study participant has known BCR-ABL-positive leukemia.
* Study participant has an active malignancy other than AML, MDS-IB2, or CMML.
* Study participant has persistent non-hematological toxicities of ≥ Grade 2 (CTCAE v4.03), with symptoms and objective findings, from prior AML, MDS-IB2, or CMML treatment (including chemotherapy, kinase inhibitors, immunotherapy, experimental agents, radiation, or surgery)
* Study participant has had hematopoietic stem cell transplant (HSCT) and meets any of the following criteria:

  1. Has undergone HSCT within the 2-month period prior to the first study dose
  2. Has clinically significant graft-versus-host-disease (GVHD) requiring treatment
  3. Has ≥ Grade 2 persistent non-hematological toxicity related to the transplant
  4. Had a donor lymphocyte infusion (DLI) ≤ 30 days prior to the first study dose.
* Study participant has meningeal or central nervous system (CNS) involvement with leukemia or other CNS disease related to underlying and secondary effects of malignancy.
* Study participant has disseminated intravascular coagulation abnormality (DIC).
* Study participant has had major surgery within 4 weeks prior to the first study dose.
* Study participant has had radiation therapy within 4 weeks prior to the first study dose.
* Study participant has congestive heart failure New York Heart Association (NYHA) class 3 or 4, or study participant with a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multigated acquisition (MUGA) scan performed within 3 months prior to study entry results in a left ventricular ejection fraction (LVEF) that is ≥ 45%.
* Study participant has any of the following cardiac abnormalities of history:

  1. Study participant has any clinically important abnormalities in rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, or PR interval > 250 milliseconds (ms).
  2. Study participant has a mean QT interval (QTc) by Friderica's method (QTcF) > 450 ms in three successive screening measurements.
  3. Study participant has any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as congenital long QT, syndrome, family history of long QT syndrome.
* Study participant is known to have active infection including any identified active COVID-19 infection.
* Study participant is known to have human immunodeficiency virus infection.
* Study participant has known active hepatitis B or C, or other active hepatic disorder.
* Study participant has any condition which, in the Investigator's opinion, makes the study participant unsuitable for study participation.
* Study participant has a history of Grade 3 or 4 non-hematologic toxicity related to tyrosine kinase inhibitor.

Inclusion Criteria for Part D:

* Study participant is defined as having morphologically documented newly diagnosed previously untreated primary or secondary AML by the World Health Organization (WHO) criteria (2016) and considered ineligible to receive intensive chemotherapy.

Study participants ≥ 75 years of age are considered ineligible to receive intensive chemotherapy if they meet any of the following criteria:

1. ECOG Performance Status of 2 or 3;
2. Cardiac history of congestive heart failure (CHF) requiring treatment or ejection fraction ≤ 50% or chronic stable angina;
3. Diffusing capacity of the lung for carbon monoxide (DLCO) ≤ 65% or forced expiratory volume during the first second (FEV1) ≤ 65%;
4. Creatinine clearance ≥ 30 mL/min to < 45 ml/min;
5. Moderate hepatic impairment with total bilirubin > 1.5 to ≤ 3.0×ULN;
6. Any other comorbidity that the Investigator judges to be incompatible with intensive chemotherapy must be reviewed and approved by the Medical Monitor during screening and prior to treatment.

Study participants are considered ineligible to receive intensive chemotherapy based on their age being ≥ 75 years.

* Study participant < 75 years has an ECOG performance status ≤ 2; study participant ≥ 75 years has an ECOG performance status 0-2.
* Study participant must meet the following criteria as indicated on the clinical laboratory tests:

  1. Serum AST and ALT ≤ 3× institutional ULN unless considered due to leukemic organ involvement.
  2. Total serum bilirubin ≤ 3x institutional ULN unless considered due to leukemic organ involvement for study participants < 75 years; total serum bilirubin ≤ 1.5x institutional ULN (or ≤ 3x institutional ULN if documented history of Gilbert's syndrome) unless considered due to leukemic organ involvement for study participants ≥ 75 years.
  3. Creatinine clearance as calculated by the Cockcroft-Gault formula or measured by 24-h urine collection of ≥ 30 mL/min for study participants < 75 years; creatinine clearance as calculated by the Cockcroft-Gault formula or measured by 24-h urine collection of ≥ 45 mL/min for study participants ≥ 75 years.
* Study participant is suitable for oral administration of study drug and has minimum life expectancy (≥ 3 months)
* Female study participants must be either:
* Of non-childbearing potential

  1. Post-menopausal (defined as at least 1 year without any menses) prior to screening, or
  2. Documented surgically sterile or status post hysterectomy (at least 1 month prior to screening)
* Or, if of childbearing potential,

  1. Must have a negative serum or urine pregnancy test at screening (within 72 hours prior to start of treatment), and
  2. Must use an acceptable highly effective contraception starting at screening and throughout the study period and for 90 days after the final study drug administration.
* Female study participants must not be breastfeeding at screening and during the study period, and for 90 days after the final study drug administration.
* Female study participants must not donate ova starting at screening and throughout the study period, and for 90 days after the final study drug administration.
* Male study participants and their female spouse/partners who are of childbearing potential must be using highly effective contraception starting at screening and continue throughout the study period and for 90 days after the final study drug administration.
* Male study participants must not donate sperm starting at screening and throughout the study period and for 90 days after the final study drug administration.
* Study participant agrees not to participate in another interventional study while on treatment.

Exclusion Criteria for Part D:

Study participants must not enter the study if any of the following exclusion criteria are met:

* Study participant was diagnosed with acute promyelocytic leukemia (APL).
* Study participant has known BCR-ABL-positive leukemia.
* Study participant has an active malignancy other than AML.
* Study participant has received treatment with the following:

  1. An HMA, VEN (or other BCL-2 inhibitor), a tyrosine kinase inhibitor (TKI), a FLT3 inhibitor (FLT3i), a hematopoietic stem cell transplant (HSCT), and/or a chemotherapeutic agent for antecedent myeloid neoplasm (Note: Prior chemotherapy for solid tumors considered in remission is allowed.)
  2. CAR-T cell therapy
  3. Experimental therapies for antecedent myeloid neoplasms
  4. Current participation in another research or observational study
* Study participant has persistent non-hematological toxicities of ≥ Grade 2 (CTCAE v4.03), with symptoms and objective findings, from treatment for antecedent myeloid neoplasms (including chemotherapy, kinase inhibitors, immunotherapy, experimental agents, immunosuppressive therapy, radiation, or surgery).
* Study participant has meningeal or central nervous system (CNS) involvement with leukemia or other CNS disease related to underlying and secondary effects of malignancy.
* Study participant has disseminated intravascular coagulation abnormality (DIC).
* Study participant has had major surgery within 4 weeks prior to the first study dose.
* Study participant has had radiation therapy within 4 weeks prior to the first study dose.
* Study participant has congestive heart failure New York Heart Association (NYHA) class 3 or 4, or study participant with a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multigated acquisition (MUGA) scan performed within 3 months prior to study entry results in a left ventricular ejection fraction (LVEF) that is ≥ 45%.
* Study participant has any of the following cardiac abnormalities of history:

  1. Study participant has any clinically important abnormalities in rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, or PR interval > 250 milliseconds (ms).
  2. Study participant has a mean QT interval (QTc) by Friderica's method (QTcF) > 450 ms in three successive screening measurements.
  3. Study participant has any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as congenital long QT, syndrome, family history of long QT syndrome.
* Study participant is known to have active infection, including any identified active COVID-19 infection.
* Study participant is known to have human immunodeficiency virus infection.
* Study participant has known active hepatitis B or C, or other active hepatic disorder.
* Study participant has any condition which, in the Investigator's opinion, makes the study participant unsuitable for study participation, including a chronic respiratory disease that requires continuous oxygen, or a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, or cardiovascular disease, or any other medical condition or known hypersensitivity to any of the study medications including excipients of VEN and AZA that in the opinion of the Investigator would adversely affect participating in this study.
* Study participant exhibits evidence of other clinically significant uncontrolled systemic infection requiring therapy (viral, bacterial, or fungal) or other medical conditions (e.g., infection, heart failure, COPD flare, etc.).
* Study participant has a white blood cell count > 25 × 10^9/L. (Treatment with hydroxyurea or use of leukapheresis are permitted to meet this criterion.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of drug-related adverse events | 4 years
Maximum tolerated dose (MTD) of tuspetinib | 4 years
  The MTD will be determined as the dose at which no more than 1 out of 6 study participants experiences a dose-limiting toxicity (DLT). Alternatively, the safety of a clinically effective dose below the MTD will be established if the MTD is not reached in study participants.
Maximum plasma concentration (Cmax) | Cycle 1 (at least 28 days)
  Maximum plasma concentration (Cmax) will be summarized by cohort using descriptive statistics including number of study participants, mean, standard deviation, minimum, median, maximum, geometric mean, and coefficient of variation (CV) of the mean and geometric mean. Time-course of drug concentrations will be plotted as appropriate.
Minimum plasma concentration (Cmin) | Cycle 1 (at least 28 days)
  Minimum plasma concentration (Cmin) will be summarized by cohort using descriptive statistics including number of study participants, mean, standard deviation, minimum, median, maximum, geometric mean, and coefficient of variation (CV) of the mean and geometric mean. Time-course of drug concentrations will be plotted as appropriate.
Area under the plasma concentration-time curve (AUC) | Cycle 1 (at least 28 days)
  Area under the plasma concentration-time curve (AUC) for various timepoints will be summarized by cohort using descriptive statistics including number of study participants, mean, standard deviation, minimum, median, maximum, geometric mean, and coefficient of variation (CV) of the mean and geometric mean. Time-course of drug concentrations will be plotted as appropriate.
Time to maximum concentration (Tmax) | Cycle 1 (at least 28 days)
  Time to maximum concentration (Tmax) will be summarized by cohort using descriptive statistics including number of study participants, mean, standard deviation, minimum, median, maximum, geometric mean, and coefficient of variation (CV) of the mean and geometric mean. Time-course of drug concentrations will be plotted as appropriate.
Terminal half-life (t1/2) | Cycle 1 (at least 28 days)
  Terminal half-life (t1/2) will be summarized by cohort using descriptive statistics including number of study participants, mean, standard deviation, minimum, median, maximum, geometric mean, and coefficient of variation (CV) of the mean and geometric mean. Time-course of drug concentrations will be plotted as appropriate.
Volume of distribution | Cycle 1 (at least 28 days)
  Volume of distribution at various timepoints will be summarized by cohort using descriptive statistics including number of study participants, mean, standard deviation, minimum, median, maximum, geometric mean, and coefficient of variation (CV) of the mean and geometric mean. Time-course of drug concentrations will be plotted as appropriate.
Plasma clearance (CL) | Cycle 1 (at least 28 days)
  Plasma clearance (CL) will be summarized by cohort using descriptive statistics including number of study participants, mean, standard deviation, minimum, median, maximum, geometric mean, and coefficient of variation (CV) of the mean and geometric mean. Time-course of drug concentrations will be plotted as appropriate.
Recommended Phase 2 dose (RP2D) of tuspetinib | 4 years
  The RP2D will be based on safety, efficacy, pharmacokinetic (PK), and pharmacodynamic (PD) considerations.

SECONDARY OUTCOMES:
Complete remission (CR) | 4 years
  Complete remission (CR) will be summarized using descriptive statistics.
Complete remission with partial hematologic recovery (CRh) | 4 years
  Complete remission with partial hematologic recovery (CRh) will be summarized using descriptive statistics.
Complete remission with incomplete platelet recovery (CRp) | 4 years
  Complete remission with incomplete platelet recovery (CRp) will be summarized using descriptive statistics.
Complete remission with incomplete hematologic recovery (CRi) | 4 years
  Complete remission with incomplete hematologic recovery (CRi) will be summarized using descriptive statistics.
Partial remission (PR) | 4 years
  Partial remission (PR) will be summarized using descriptive statistics.
Overall response rate | 4 years
  Overall response rate will be summarized using descriptive statistics.
Duration of response | 4 years
  Survival curves and median for time-to-event variables will be estimated using the Kaplan-Meier method and will be reported along with corresponding 95% confidence intervals.
Disease-free survival (DFS) | 4 years
  Survival curves and median for time-to-event variables will be estimated using the Kaplan-Meier method and will be reported along with corresponding 95% confidence intervals.
Overall survival (OS) | 4 years
  Survival curves and median for time-to-event variables will be estimated using the Kaplan-Meier method and will be reported along with corresponding 95% confidence intervals.
Event-free survival (EFS) | 4 years
  Survival curves and median for time-to-event variables will be estimated using the Kaplan-Meier method and will be reported along with corresponding 95% confidence intervals.

OTHER OUTCOMES:
Percent inhibition of phosphorylation of targeted proteins | 4 years
  Flow cytometry will be used to identify leukemic blasts and quantify levels of phosphorylated targeted proteins including FLT3 and STAT5, among others, using a plasma inhibitory activity (PIA) assay that exposes cell lines to plasma from study participants treated in the study.
Mutation status of genes after treatment with tuspetinib | 4 years
  Mutation status of genes including, but limited to, FLT3, NRAS, and TP53

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (34):
- United States (15):
  - The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Irvine, Irvine, California
  - UCSD Moores Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - University of California, Davis, Sacramento, California
  - Yale University, New Haven, Connecticut
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic - Taussig Cancer Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - MD Anderson Cancer Center, Huston, Texas
- Australia (5):
  - Border Medical Oncology, Albury, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Townsville University Hospital, Townsville, Queensland
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Germany (2):
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Charité Universitätsmedizin Berlin, Berlin, State of Berlin
- Auckland City Hospital, Grafton, Auckland, New Zealand
- South Korea (6):
  - Seoul National University Hospital, Seoul, Seoul
  - Asan Medical Center, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
  - Kyungpook National University Hospital, Daegu
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
- Spain (5):
  - Hospital Universitario Vall d'Hebron, Barcelona, Barcelona
  - Hospital Quirón Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia, Valencia

REFERENCES:
- [Derived] Sonowal H, Rice WG, Bejar R, Byun JY, Jung SH, Sinha R, Howell SB. Preclinical Development of Tuspetinib for the Treatment of Acute Myeloid Leukemia. Cancer Res Commun. 2025 Jan 1;5(1):74-83. doi: 10.1158/2767-9764.CRC-24-0258. PMID 39665627